CLINICAL TRIAL: NCT02796781
Title: Autologous Lung Stem Cell Transplantation in Patients With Interstitial Lung Diseases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Regend Therapeutics (Industry)
Responsible Party: Principal Investigator, Wei Zuo, Professor, Shanghai East Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201602102
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Interstitial Lung Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lung stem cells (Experimental): Patients will receive 0.5-5x10^6 (0.5-5 million)/Kg/person cells of clinical grade lung stem cells (LSCs)injected into lung via fiberoptic bronchoscopy.
  Interventions: Biological: Lung stem cells

INTERVENTIONS:
Biological: Lung stem cells — Patients will receive clinical grade lung stem cells (LSCs)injected into lung via fiberoptic bronchoscopy.

SUMMARY:
Interstitial lung diseases (ILD) are a group of diseases affecting the lung interstitium. The lung scarring that occurs in ILD is often irreversible with only mitigating therapy available so far. This study intends to carry out an open, single-armed, phase I/II clinical trial to investigate whether lung stem cells can regenerate damaged lung tissue. During the treatment, lung stem cells will be isolated from patients' own bronchi and expanded in vitro. After careful characterization, cultured cells will be injected directly into the lesion by fiberoptic bronchoscopy. The safety and efficacy of the treatment will be monitored by measuring the key clinical indicators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with interstitial lung disease
* Clinically stable
* Written informed consent signed

Exclusion Criteria:

* Allergic to cell therapy;
* Patients with serious significant pulmonary infection need anti-infection treatment;
* Patients who has taken amiodarone which may cause pulmonary fibrosis in the past 3 months;
* Patients with malignant tumor in the past 5 years;
* Participated in other clinical trials in the past 3 months;
* Patients with serious heart disease(NYHA class Ⅲ-Ⅳ)
* Pregnant or lactating women;
* The investigator assessed as inappropriate to participate in this clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Increase of diffusing capacity of the lung for carbon monoxide (DLCO) | 24 weeks

SECONDARY OUTCOMES:
Increase of total lung capacity (TLC) | 24 weeks
Increase in 6 minute walk distance (6MWD) | 24 weeks
Life quality: assessed by St. George respiratory questionnaire (SGRQ) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuo W, Zhang T, Wu DZ, Guan SP, Liew AA, Yamamoto Y, Wang X, Lim SJ, Vincent M, Lessard M, Crum CP, Xian W, McKeon F. p63(+)Krt5(+) distal airway stem cells are essential for lung regeneration. Nature. 2015 Jan 29;517(7536):616-20. doi: 10.1038/nature13903. Epub 2014 Nov 12. PMID 25383540